CLINICAL TRIAL: NCT00765817
Title: A Randomized Trial Comparing Exenatide With Placebo in Subjects With Type 2 Diabetes on Insulin Glargine With or Without Oral Antihyperglycemic Medications
Brief Title: Addition Of Exenatide To Insulin Glargine In Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-US-GWCO
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; exenatide; Amylin; Lilly; metformin; pioglitazone; insulin glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental)
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: placebo — subcutaneous injection, twice a day
  Arms: 1
Drug: exenatide — subcutaneous injection, twice a day, 10mcg
  Arms: 2

SUMMARY:
This study will compare the efficacy and safety of exenatide versus placebo in adults whose diabetes is not fully controlled by insulin glargine with or without metformin and/or pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes.
* Have been taking insulin glargine at a dose of ≥20 units/day for at least 3 months before entering the study.

Have been taking insulin glargine alone or in combination with one of the following for at least 3 months before entering the study:

1. metformin (stable dose for 6 weeks)
2. pioglitazone (stable dose for 6 weeks)
3. a combination of metformin and pioglitazone (stable dose for 6 weeks)

   * Have HbA1C between 7.1% and 10.5%, inclusive.
   * Have a body mass index (BMI) ≤45 kg/m2.
   * Have a history of stable body weight (not varying by >5% for at least 3 months prior to screening).

Exclusion Criteria:

* Have taken medications to lower blood sugar other than insulin glargine, pioglitazone, or metformin in the 3 months before entering the study for more than a 1-week period, or within 1 week of entering the study.
* Have had more than one episode of major (severe) hypoglycemia in the 6 months before entering the study.
* Are pregnant or intend to become pregnant during the study or are sexually active women not actively practicing birth control.
* Women who are breastfeeding.
* Have any significant diseases of the blood, heart, kidney, gastrointestinal system, or other significant diseases such as cancer.
* Have had a kidney transplant or are currently on kidney dialysis.
* Have a cancer that's never been treated, that's currently being treated, or that was diagnosed within the last 5 years.
* Have had a bad reaction to exenatide in the past or have a condition that is not recommended to be exposed to exenatide or any of exenatide's other ingredients.
* Have used a drug for weight loss in the 3 months before entering the study for more than a 1-week period, or within 1 month of entering the study.
* Are currently on a weight-loss program or have been on one within 3 months of entering the study.
* Have had a blood transfusion or severe blood loss within 3 months of entering the study.
* Are taking systemic glucocorticoids or have received systemic glucocorticoids within 8 weeks of entering the study.
* Have an irregular sleep cycle (for example, sleeping during the day and working during the night).
* Have a history of pancreatitis.
* Have received treatment with an experimental drug within 30 days of entering the study.
* If on metformin, have a condition that is not recommended to be exposed to metformin, or any condition associated with hypoperfusion, hypoxemia, dehydration, or sepsis.
* If on metformin, have had a radiologic contrast study performed within 48 hours of entering the study.
* If on pioglitazone, have a condition that is not recommended to be exposed to pioglitazone, including congestive heart failure, or are taking pioglitazone at a dose that is not approved for use with insulin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (59):
- United States (40):
  - Research Site, Peoria, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Buena Park, California
  - Research Site, Concord, California
  - Research Site, Fresno, California
  - Research Site, Greenbrae, California
  - Research Site, La Mesa, California
  - Research Site, Lancaster, California
  - Research Site, Northridge, California
  - Research Site, Palm Springs, California
  - Research Site, Salinas, California
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Idaho Falls, Idaho
  - Research Site, Des Moines, Iowa
  - Research Site, Wichita, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Matairie, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Chesterfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Berkeley Heights, New Jersey
  - Research SIte, Teaneck, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research SIte, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Bend, Oregon
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Georgetown, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Vancouver, Washington
  - Research Site, Kenosha, Wisconsin
- Greece (2):
  - Research Site, Athens, Greece
  - Research Site, Thessaloniki, Greece
- Israel (3):
  - Research Site, Holon, Israel
  - Research Site, Kfar Saba, Israel
  - Research Site, Tel Litwinsky, Israel
- Mexico (3):
  - Research Site, Coatzacoalcos, Mexico
  - Research Site, Monterrey, Mexico
  - Research Site, México, State of Mexico
- Puerto Rico (4):
  - Research Site, Carolina
  - Research Site, Hato Rey
  - Research Site, Ponce
  - Research Site, San Juan
- United Kingdom (7):
  - Research Site, Birmingham, United Kingdom
  - Research Site, Guildford, United Kingdom
  - Research Site, Leicester, United Kingdom
  - Research Site, Livingston, United Kingdom
  - Research Site, Middlesbrough, United Kingdom
  - Research Site, Swansea, United Kingdom
  - Research Site, Torquay, United Kingdom

REFERENCES:
- [Derived] Buse JB, Han J, Miller S, MacConell L, Pencek R, Wintle M. Addition of exenatide BID to insulin glargine: a post-hoc analysis of the effect on glycemia and weight across a range of insulin titration. Curr Med Res Opin. 2014 Jul;30(7):1209-18. doi: 10.1185/03007995.2014.896329. Epub 2014 Mar 18. PMID 24621255
- [Derived] Zinman B, Philis-Tsimikas A, Cariou B, Handelsman Y, Rodbard HW, Johansen T, Endahl L, Mathieu C; NN1250-3579 (BEGIN Once Long) Trial Investigators. Insulin degludec versus insulin glargine in insulin-naive patients with type 2 diabetes: a 1-year, randomized, treat-to-target trial (BEGIN Once Long). Diabetes Care. 2012 Dec;35(12):2464-71. doi: 10.2337/dc12-1205. Epub 2012 Oct 5. PMID 23043166
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891
- [Derived] Rosenstock J, Shenouda SK, Bergenstal RM, Buse JB, Glass LC, Heilmann CR, Kwan AY, MacConell LA, Hoogwerf BJ. Baseline factors associated with glycemic control and weight loss when exenatide twice daily is added to optimized insulin glargine in patients with type 2 diabetes. Diabetes Care. 2012 May;35(5):955-8. doi: 10.2337/dc11-1434. Epub 2012 Mar 19. PMID 22432107
- [Derived] Buse JB, Bergenstal RM, Glass LC, Heilmann CR, Lewis MS, Kwan AY, Hoogwerf BJ, Rosenstock J. Use of twice-daily exenatide in Basal insulin-treated patients with type 2 diabetes: a randomized, controlled trial. Ann Intern Med. 2011 Jan 18;154(2):103-12. doi: 10.7326/0003-4819-154-2-201101180-00300. Epub 2010 Dec 6. PMID 21138825

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects who started the study, subsequently withdrew prior to receiving study medication and are not part of the full analysis set
Groups:
- Exenatide Arm: Exenatide 5mcg twice daily for 4 weeks, followed by exenatide 10mcg twice daily for 26 weeks (with a background of titrated insulin glargine and other oral antidiabetic agents)
- Placebo Arm: Placebo volume equivalent to the active volume injected in the exenatide arm (with a background of titrated insulin glargine and other oral antidiabetic agents)
Period: Overall Study
Arm/Group | Exenatide Arm | Placebo Arm
Started | 138 (One subject withdrew prior to receiving study medication, not included in analysis set) | 123 (One subject withdrew prior to receiving study medication, not included in analysis set)
Completed | 112 | 101
Not Completed | 26 | 22
Not completed — Adverse Event | 13 | 1
Not completed — Death | 0 | 1
Not completed — Entry criteria not met | 2 | 2
Not completed — Loss of glucose control | 0 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Subject decision | 7 | 11

BASELINE CHARACTERISTICS:
Population: One subject per group withdrew from the study prior to the first dose of study medication and therefore are not part of the baseline or subsequent analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Arm | Placebo Arm | Total
Number analyzed (Participants) | 137 | 122 | 259
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 84 | 184
  >=65 years | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.67 (8.91) | 59.40 (9.96) | 59.01 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 44 | 111
  Male | 70 | 78 | 148

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c)
Description: Change in HbA1c from baseline following 30 weeks of therapy (i.e., HbA1c at week 30 minus HbA1c at baseline). Unit of measure is percent of hemoglobin that is glycosylated.
Time Frame: baseline and 30 weeks
Population: Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 112 | 100
percentage of hemoglobin | -1.71 (0.09) | -1.00 (0.09)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Secondary Outcome: Percentage of Patients Achieving HbA1c <=7%
Description: Percentage of patients in each arm who had HbA1c >7% at baseline and had HbA1c <=7% at week 30 (percentage = [number of subjects with HbA1c <=7% at week 30 divided by number of subjects with HbA1c >7% at baseline] * 100%).
Time Frame: baseline and 30 weeks
Population: Full analysis set. Last observation carried forward. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis. Only patients with baseline HbA1c > target were included in calculation.
Measure: Number; unit: percentage
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 127 | 106
percentage | 58.3 | 31.1
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Patients Achieving HbA1c <=6.5%
Description: Percentage of patients in each arm who had HbA1c >6.5% at baseline and had HbA1c <=6.5% at week 30 (percentage = [number of subjects with HbA1c <=6.5% at week 30 divided by number of subjects with HbA1c >6.5% at baseline] * 100%).
Time Frame: baseline and 30 weeks
Population: as for outcome 2
Measure: Number; unit: percentage
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 131 | 113
percentage | 42.0 | 13.3
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Change in Fasting Serum Glucose
Description: Change in fasting serum glucose following 30 weeks of therapy (i.e., fasting serum glucose at week 30 minus fasting serum glucose at baseline)
Time Frame: baseline and 30 weeks
Population: Full analysis set, Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 111 | 98
mmol/L | -1.28 (0.2) | -0.87 (0.2)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.174, ANCOVA

5. Secondary Outcome: Change in 7-point Self-monitored Blood Glucose (SMBG) Profile
Description: Change in 7-point (pre-breakfast, 2 hour post-breakfast, pre-lunch, 2 hour post-lunch, pre-dinner, 2 hour post-dinner, 0300 hours) SMBG profile from baseline to week 30 (change = blood glucose value at week 30 minus blood glucose value at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 108 | 89
mmol/L
  Pre-breakfast: baseline | 7.89 (0.2) | 8.27 (0.2)
  Pre-breakfast: change at week 30 | -1.58 (0.1) | -1.48 (0.1)
  2 hour post-breakfast: baseline | 10.89 (0.2) | 11.82 (0.2)
  2 hour post-breakfast: change at week 30 | -3.56 (0.2) | -1.72 (0.2)
  Pre-lunch: baseline | 8.95 (0.2) | 9.77 (0.2)
  Pre-lunch: change at week 30 | -2.23 (0.2) | -1.15 (0.2)
  2 hour post-lunch: baseline | 11.35 (0.2) | 11.70 (0.2)
  2 hour post-lunch: change at week 30 | -2.74 (0.2) | -1.38 (0.2)
  Pre-dinner: baseline | 9.85 (0.2) | 9.99 (0.2)
  Pre-dinner: change at week 30 | -2.25 (0.2) | -1.33 (0.2)
  2 hour post-dinner: baseline | 12.03 (0.3) | 11.86 (0.3)
  2 hour post-dinner: change at week 30 | -3.87 (0.2) | -1.34 (0.3)
  0300: baseline | 8.95 (0.2) | 9.20 (0.2)
  0300: change at week 30 | -2.27 (0.2) | -1.48 (0.2)

6. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol following 30 weeks of therapy (i.e., total cholesterol at week 30 minus total cholesterol at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 110 | 98
mmol/L | -0.16 (0.08) | -0.02 (0.09)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.203, ANCOVA

7. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol
Description: Change in LDL cholesterol following 30 weeks of therapy (i.e., LDL cholesterol at week 30 minus LDL cholesterol at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 102 | 97
mmol/L | -0.19 (0.07) | -0.00 (0.07)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.063, ANCOVA

8. Secondary Outcome: Change in High Density Lipoprotein (HDL) Cholesterol
Description: Change in HDL cholesterol following 30 weeks of therapy (i.e., HDL cholesterol at week 30 minus HDL cholesterol at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 110 | 98
mmol/L | 0.01 (0.02) | 0.00 (0.02)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.745, ANCOVA

9. Secondary Outcome: Change in Triglycerides
Description: Change in triglycerides following 30 weeks of therapy (i.e., triglycerides at week 30 minus triglycerides at baseline)
Time Frame: baseline and 30 weeks
Population: Full analysis set. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 110 | 98
mmol/L | -0.02 (0.09) | -0.03 (0.09)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.933, ANCOVA

10. Secondary Outcome: Change in Body Weight
Description: Change in body weight following 30 weeks of therapy (i.e., body weight at week 30 minus body weight at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 112 | 101
kg | -1.78 (0.3) | 0.96 (0.3)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p < 0.001, ANCOVA

11. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference following 30 weeks of therapy (i.e., waist circumference at week 30 minus waist circumference at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 137 | 120
cm | -1.08 (0.52) | -0.25 (0.55)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.226, ANCOVA

12. Secondary Outcome: Change in Daily Insulin Dose
Description: Change in daily insulin dose following 30 weeks of therapy (i.e., daily insulin dose at week 30 minus daily insulin dose at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: insulin units (U)
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 110 | 100
insulin units (U) | 13.19 (2.02) | 19.71 (2.11)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.026, ANCOVA

13. Secondary Outcome: Change in Daily Insulin Dose (on a Per Body Weight Basis)
Description: Change in daily insulin dose per kilogram (kg) following 30 weeks of therapy (i.e., daily insulin dose per kg at week 30 minus daily insulin dose per kg at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: insulin units per kg (U/kg)
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 110 | 100
insulin units per kg (U/kg) | 0.15 (0.02) | 0.20 (0.02)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.070, ANCOVA

14. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change in SBP following 30 weeks of therapy (i.e., SBP at week 30 minus SBP at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 112 | 101
mmHg | -2.74 (1.2) | 1.71 (1.3)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.011, ANCOVA

15. Secondary Outcome: Change in Diastolic Blood Pressure (DBP)
Description: Change in DBP following 30 weeks of therapy (i.e., DBP at week 30 minus DBP at baseline)
Time Frame: baseline and 30 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 112 | 101
mmHg | -1.73 (0.6) | 1.69 (0.7)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p < 0.001, ANCOVA

16. Secondary Outcome: Minor Hypoglycemia Rate Per Year
Description: Number of minor hypoglycemia events experienced per subject per year. Minor hypoglycemia was defined as any time a subject felt he or she was experiencing a sign or symptom associated with hypoglycemia that was either self-treated by the subject or resolved on its own and had a concurrent finger stick blood glucose <3.0 mmol/L (54 mg/dL).
Time Frame: baseline and weeks 2, 4, 6, 8, 10, 14, 18, 22, 26, and 30
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: events per subject per year
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 137 | 122
events per subject per year | 1.61 (5.94) | 1.55 (4.79)
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.666, Negative binomial regression model

17. Secondary Outcome: Percentage of Subjects Experiencing Minor Hypoglycemia
Description: Percentage of subjects in each arm experiencing at least one episode of minor hypoglycemia at any point during the study. Minor hypoglycemia was defined as any time a subject felt he or she was experiencing a sign or symptom associated with hypoglycemia that was either self-treated by the subject or resolved on its own and had a concurrent finger stick blood glucose <3.0 mmol/L (54 mg/dL).
Time Frame: baseline and weeks 2, 4, 6, 8, 10, 14, 18, 22, 26, and 30
Population: Full analysis set
Measure: Number; unit: percentage
Arm/Group | Exenatide Arm | Placebo Arm
Number analyzed (Participants) | 137 | 122
percentage | 24.8 | 28.7
Statistical Analysis 1: Comparison: Exenatide Arm vs Placebo Arm; Test type: Superiority or Other; p = 0.486, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Exenatide Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 8/137 | 11/122
Other Adverse Events (participants affected / at risk) | 109/138 | 66/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Arm (N=137) | Placebo Arm (N=122)
Chest pain (General disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eye penetration (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Small intestine obstruction (Gastrointestinal disorders) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Transient ischemic attack (Cardiac disorders) | 0 | 1
Uticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Arm (N=138) | Placebo Arm (N=123)
Nausea (Gastrointestinal disorders) | 56 | 10
Diarrhea (Gastrointestinal disorders) | 25 | 10
Vomiting (Gastrointestinal disorders) | 25 | 5
Headache (Nervous system disorders) | 19 | 5
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Constipation (Gastrointestinal disorders) | 14 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Nasopharyngitis (Infections and infestations) | 8 | 6
Dizziness (Nervous system disorders) | 6 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 2
Dyspepsia (Gastrointestinal disorders) | 9 | 2
Asthenia (General disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days